CLINICAL TRIAL: NCT02557100
Title: A Randomized, Head-to-Head, Single-Blinded Study to Assess Changes in the Immune Profile in Response to Treatment With Subcutaneous Abatacept in Combination With Methotrexate Versus Subcutaneous Adalimumab in Combination With Methotrexate in Adults With Early Rheumatoid Arthritis Who Are Naive to Biologic Disease-Modifying Antirheumatic Drugs
Brief Title: Study to Assess Changes in the Immune Profile in Adults With Early Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IM101-567
Record Dates: First submitted 2015-09-04; First posted 2015-09-23 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Adalimumab; Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Abatacept Single Blind Treatment Period
  Interventions: Drug: Abatacept; Drug: Methotrexate
- Treatment B (Active Comparator): Adalimumab Single Blind Treatment Period
  Interventions: Drug: Abatacept; Drug: Adalimumab; Drug: Methotrexate
- Treatment C (Active Comparator): Abatacept Cumulative Treatment Period
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept
  Other Names: Orencia
Drug: Adalimumab
  Other Names: Humira
  Arms: Treatment B
Drug: Methotrexate
  Arms: Treatment A; Treatment B

SUMMARY:
The purpose of this study is to examine changes in immune cells and proteins in response to treatment with two approved therapies for Rheumatoid arthritis (RA), abatacept versus adalimumab, both given in combination with methotrexate.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Symptoms of RA for no more than 12 months prior to enrollment
* Meet American College of Rheumatology/European League against Rheumatism (ACR/EULAR) 2010 criteria for classification of RA
* Treated with Methotrexate (MTX) for at least 12 weeks prior to randomization with a stable oral dose for at least 4 weeks, Subjects must randomize on the maximum tolerated dose of oral methotrexate (minimum of 15 mg and maximum of 25 mg per week), dose of MTX < 15 mg/week but ≥ 7.5 mg/week is permitted if subjects are intolerant to higher doses
* At least 3 tender & 3 swollen joints
* Anti-cyclic citrullinated peptide (CCP) > 3X the upper limit of normal and positive rheumatoid factor

Exclusion Criteria:

* History of other autoimmune diseases (eg, psoriasis, systemic lupus, erythematosus, etc)
* Prior use of non-biologic therapy other than methotrexate
* Prior use of biologic and targeted synthetic disease-modifying anti-rheumatic drugs (DMARD) therapy
* Subjects with chronic or recent acute serious infection

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (28):
- United States (21):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Rheumatology Associates Of North Alabama, P.C., Huntsville, Alabama
  - Clinical And Translational Research Center Of Alabama, Pc, Tuscaloosa, Alabama
  - Arizona Arthritis & Rheumatology Research PLLC, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research PLLC, Phoenix, Arizona
  - St. Joseph Heritage Medical Group, Fullerton, California
  - Desert Medical Advances, Palm Desert, California
  - University Of Colorado Health Sciences Center, Aurora, Colorado
  - Medical Faculty Associates,Inc., Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Integral Rheumatology & Immunology Specialists, Plantation, Florida
  - Marietta Rheumatology, Marietta, Georgia
  - The Center For Rheumatology And Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Aa Mrc Llc, Grand Blanc, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Oregon Health & Science University (Ohsu), Portland, Oregon
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Carolina Health Specialists, Myrtle Beach, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Arthritis Clinic Of Northern Virginia, P.C., Arlington, Virginia
- Canada (4):
  - Dr. Anil K Gupta Med Prof Corp, Toronto, Ontario
  - Essex County Medical Society, Windsor, Ontario
  - Institut De Rhumatologie De Montreal, Montreal, Quebec
  - Centre De Recherche Musculo-Squelettique, Trois-Rivières, Quebec
- Mexico (3):
  - Clinica de Investigacion en Reumatologia y Obesidad S.C., Guadalajara, Jalisco
  - CINTRE - Centro de investigacion y tratamiento reumatologico, S.C., Mexico City, Mexico City
  - Clinica Integral en Osteoporosis y Artritis CLINOSAR Mexico S.A. de C.V., Mexico City

REFERENCES:
- [Derived] Rigby W, Buckner JH, Louis Bridges S Jr, Nys M, Gao S, Polinsky M, Ray N, Bykerk V. HLA-DRB1 risk alleles for RA are associated with differential clinical responsiveness to abatacept and adalimumab: data from a head-to-head, randomized, single-blind study in autoantibody-positive early RA. Arthritis Res Ther. 2021 Sep 18;23(1):245. doi: 10.1186/s13075-021-02607-7. PMID 34537057
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 80 participants randomized and treated.
Groups:
- Treatment C: Cumulative Abatacept Period
Period: Single Blind Treatment Period
Arm/Group | Treatment A | Treatment B | Treatment C
Started (= treated) | 40 | 40 | 0
Completed (= completed treatment) | 40 | 36 | 0
Not Completed | 0 | 4 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Request to Discontinue | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Transition to Open Label
Arm/Group | Treatment A | Treatment B | Treatment C
Started | 40 | 36 | 0
Completed | 0 | 0 | 0
Not Completed | 40 | 36 | 0
Not completed — Entered Cumulative Abatacept Period | 40 | 36 | 0
Period: Cumulative Abatacept Period
Arm/Group | Treatment A | Treatment B | Treatment C
Started | 0 | 0 | 76
Completed | 0 | 0 | 72
Not Completed | 0 | 0 | 4
Not completed — Other Reasons | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Request to Discontinue | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Participants treated in the single-blind period
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Treatment C | Total
Number analyzed (Participants) | 40 | 40 | 0 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.2 (12.16) | 44.7 (16.30) |  | 46.0 (14.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 |  | 60
  Male | 11 | 9 |  | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 |  | 10
  Not Hispanic or Latino | 16 | 14 |  | 30
  Unknown or Not Reported | 20 | 20 |  | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 2 |  | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 4 | 1 |  | 5
  White | 36 | 36 |  | 72
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Adverse Events (AEs)
Description: Percentage of participants who experienced an AE
Time Frame: up to 85 days post last dose, approximately 40 weeks
Population: All Treated Participants
Measure: Number; unit: Percentage of participant with AEs
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 40 | 40 | 76
Percentage of participant with AEs | 55.0 | 70.0 | 57.9

2. Primary Outcome: Percentage of Participants With an Serious Adverse Events (SAEs)
Description: Percentage of participants who experienced an SAEs
Time Frame: up to 85 days post last dose, approximately 40 weeks
Population: All treated participants
Measure: Number; unit: Percentage of participants with SAEs
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 40 | 40 | 76
Percentage of participants with SAEs | 2.5 | 5.0 | 5.3

3. Primary Outcome: Percentage of Participants With Adverse Events Leading to Discontinuation (AEsDc)
Description: Percentage of participants who experienced an (AEsDc)
Time Frame: up to 85 days post last dose, approximately 40 weeks
Population: All Treated Participants
Measure: Number; unit: Percentage of participants with AEsDC
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 40 | 40 | 76
Percentage of participants with AEsDC | 0 | 2.5 | 0

4. Primary Outcome: Percentage of Serious Adverse Events Leading to Discontinuation (SAEsDc)
Description: Percentage of participants who experienced an (SAEsDc)
Time Frame: up to 85 days post last dose, approximately 40 weeks
Population: All Treated Participants
Measure: Number; unit: Percentage of participants with SAEsDc
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 40 | 40 | 76
Percentage of participants with SAEsDc | 0 | 2.5 | 0

5. Primary Outcome: Percentage of Drug Related Adverse Events (DRAEs)
Description: Percentage of participants who experienced an DRAEs
Time Frame: up to 85 days post last dose, approximately 40 weeks
Population: All Treated Participants
Measure: Number; unit: Percentage of participants with DRAEs
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 40 | 40 | 76
Percentage of participants with DRAEs | 30.0 | 27.5 | 22.4

6. Primary Outcome: Percentage of Drug Related Serious Adverse Events (DRSAEs)
Description: Percentage of participants who experienced an DRSAEs
Time Frame: up to 85 days post last dose, approximately 40 weeks
Population: All Treated Participants
Measure: Number; unit: Percentage of Participants with DRSAEs
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 40 | 40 | 76
Percentage of Participants with DRSAEs | 0 | 2.5 | 0

7. Primary Outcome: Number of Deaths
Description: Number of participants who experienced Death
Time Frame: up to 85 days post last dose, approximately 40 weeks
Population: All Treated Participants
Measure: Number; unit: Number of Deaths
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 40 | 40 | 76
Number of Deaths | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: up to 85 days post last dose, approximately 40 weeks
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 0/40 | 1/40 | 0/76
Serious Adverse Events (participants affected / at risk) | 1/40 | 2/40 | 4/76
Other Adverse Events (participants affected / at risk) | 21/40 | 28/40 | 19/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=40) | Treatment B (N=40) | Treatment C (N=76)
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 | 0 | 1
Sudden Death (General disorders) | 0 | 1 | 0
Varicella (Infections and infestations) | 0 | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 1
Incision site complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=40) | Treatment B (N=40) | Treatment C (N=76)
Upper respiratory tract infection (Infections and infestations) | 3 | 14 | 10
Nasopharyngitis (Infections and infestations) | 4 | 2 | 5
Urinary Tract Infection (Infections and infestations) | 4 | 0 | 5
Alanine Aminotransferase Increased (Investigations) | 3 | 6 | 9
Aspartate Aminotransferase Increased (Investigations) | 2 | 5 | 7
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 2
Headache (Nervous system disorders) | 2 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2015-07-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT02557100/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT02557100/SAP_001.pdf